CLINICAL TRIAL: NCT04233164
Title: Genomic Effects of Glucocorticoids in Patients With Systemic Lupus Erythematosus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 200032; 20-AR-0032
Record Dates: First submitted 2020-01-16; First posted 2020-01-18 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-03

CONDITIONS: Systemic Lupus Erythematous (SLE)
Keywords: Immunosuppressive Drugs; Methylprednisolone; PREDNISONE; Steroids; Autoimmunity
MeSH Terms: conditions — Autoimmune Diseases | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Glucocorticoids 1 mg/kg dose (Experimental): Participants with Systemic Lupus Erythematosus (SLE) received a single intravenous dose of methylprednisolone 1 mg/kg and blood was collected two hours and four hours after the start of the infusion.
  Interventions: Drug: Solu-Medrol 1mg/kg
- Group B: Glucocorticoids 250 mg dose (Experimental): Participants with Systemic Lupus Erythematosus (SLE) received a single intravenous dose of 250 mg of methylprednisolone and blood was collected two hours and four hours after the start of the infusion.
  Interventions: Drug: Solu-Medrol 250 mg

INTERVENTIONS:
Drug: Solu-Medrol 1mg/kg — Methylprednisolone sodium succinate for injection, United States Pharmacopeia grade (USP), sold as SOLU-MEDROL sterile powder by Pfizer, Inc, is an anti-inflammatory glucocorticoid that occurs as a white, or nearly white, odorless hygroscopic, amorphous solid. It is very soluble in water and in alcohol, but is insoluble in chloroform and is very slightly soluble in acetone. The study agent solution will be administered as an IV infusion over 30 minutes, for a total single dose of 1 mg/kg of methylprednisolone.
  Arms: Group A: Glucocorticoids 1 mg/kg dose
Drug: Solu-Medrol 250 mg — Methylprednisolone sodium succinate for injection, United States Pharmacopeia grade (USP), sold as SOLU-MEDROL sterile powder by Pfizer, Inc, is an anti-inflammatory glucocorticoid that occurs as a white, or nearly white, odorless hygroscopic, amorphous solid. It is very soluble in water and in alcohol, but is insoluble in chloroform and is very slightly soluble in acetone. The study agent solution will be administered as an IV infusion over 30 minutes, for a total single dose of 250 mg of methylprednisolone.
  Arms: Group B: Glucocorticoids 250 mg dose

SUMMARY:
Background:

The immune system is the body's defense against bacteria and other harmful invaders. In people with systemic lupus erythematosus (SLE), the immune system becomes overactive and attacks healthy cells by mistake. Many people use glucocorticoids (GCs) to treat their SLE. GCs can calm down an overactive immune system by changing how the body reads genes. But GCs have side effects that can increase over time. Researchers want to learn more about how GCs work. This may help to develop new and better drugs for treating SLE without the side effects GCs have.

Objective:

To better understand how GCs affect the immune system in people with SLE.

Eligibility:

People age 18-80 with SLE.

Design:

Participants will be screened with a physical exam. They will have a health and medical history. They will have blood and urine tests. They will have an electrocardiogram to measure heart activity. For this, sticky pads are put on their chest, arms, and legs.

Participants will have a methylprednisolone infusion for about 30 minutes. It will be given through a needle in a vein.

Blood will be collected immediately before, 2 hours after, and 4 hours after the start of the infusion. Blood pressure and heart activity will be monitored. Participants will repeat some of the screening tests.

Participants will be contacted twice in the week after the infusion visit. They will discuss any health problems they are having.

DETAILED DESCRIPTION:
Study Design:

This is a study of the acute effects of glucocorticoids on the immune system of patients with SLE. Participants will undergo baseline blood collection prior to receiving a single intravenous (IV) dose of methylprednisolone sodium succinate. Participants will be randomized into 1 of 2 dose groups: 1 mg/kg or 250 mg. Blood will be collected again at 2 and 4 hours after the methylprednisolone infusion. Individual participation requires 2 visits to the NIH CC and 2 follow-up phone calls. Total length of individual subject participation including screening is 1-12 weeks. Blood samples will be processed for isolation of hematopoietic cell sub-populations (eg, neutrophils, B cells, plasmacytoid dendritic cells, CD4+ T cells, CD8+ T cells, monocytes, and natural killer cells). Laboratory studies will be performed on the purified cells, with the goal of understanding the human response to glucocorticoids in vivo at the level of circulating cell populations (eg, flow cytometry, mass cytometry), RNA (eg, RNA sequencing [RNA-seq], small-RNA-seq, real-time polymerase chain reaction [PCR]), DNA (eg, chromatin immunoprecipitation sequencing [ChIP-seq], methylation analysis, DNA sequencing, genotyping), and protein (eg, flow cytometry, mass spectrometry). At each time point, serum methylprednisolone levels will be measured.

Study Agent/ Intervention Description:

A single IV infusion of methylprednisolone sodium succinate at either 1 mg/kg or 250 mg.

Primary Objective:

To understand the cellular and molecular response to glucocorticoids in individuals with SLE.

Glucocorticoid Genomics in SLE

Secondary Objectives:

1. To identify candidate targets for therapeutic interventions that could mimic the action of glucocorticoids in patients with SLE, without the significant toxicity caused by the broad range of glucocorticoid actions.
2. To test whether the transcriptional response to glucocorticoids differs between the two doses being studied.
3. To identify similarities and differences, at baseline and in response to glucocorticoids, between the transcriptome of cells from patients and those from the previously studied healthy subjects.

Primary Endpoint:

A list of human protein-coding genes and non-coding RNAs that are differentially expressed in response to glucocorticoids in patients with SLE, for each of the studied cell types and doses.

Secondary Endpoints:

1. A comparison of the transcriptional response to glucocorticoids between the two dose groups.
2. A list of protein-coding and non-coding transcripts, their corresponding proteins, and the molecular pathways representing the best candidates for targeted therapeutic alternatives to glucocorticoids.
3. Validation of the targets identified by functional studies.
4. For each cell type, a list of protein-coding or non-coding transcripts that are shared and a list of transcripts that are different, between patients with SLE and the previously studied healthy controls, at baseline or in response to glucocorticoids.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Aged 18-80 years.
  2. Has a diagnosis of SLE based on the 1997 Update of the 1982 American College of Rheumatology Revised Criteria for Classification of SLE.
  3. Currently enrolled in study 94-AR-0066.
  4. Able to provide informed consent.
  5. Willing to allow genetic testing.
  6. Has a primary care physician or other healthcare provider who will manage all health conditions related or unrelated to the study objectives.
  7. If receiving immunosuppressive therapies other than glucocorticoids for SLE, then on a stable dose (defined as no increases in dose for the 60 days prior to screening).
  8. A. If receiving glucocorticoid therapy and not experiencing a lupus flare at the time of the screening visit, then potential participants must be on a daily prednisone or prednisone-equivalent dose less than or equal to 10 mg/day and agree to undergo a glucocorticoid taper.

B. If receiving glucocorticoid therapy experiencing a lupus flare at the time of the screening visit, then potential participants must be on a daily prednisone or prednisone-equivalent dose less than or equal to 15mg/day. A glucocorticoid taper will not be performed.

EXCLUSION CRITERIA:

1. Body mass index (BMI) < 18 or > 40.
2. History of a severe allergic reaction to glucocorticoids.
3. History of a severe adverse cardiovascular or psychiatric event related to glucocorticoid administration.
4. Use of a glucocorticoid at a prednisone-equivalent dose 10 mg/day in the 15 days prior to screening (> 15 mg/day if experiencing a flare on the day of the screening visit).
5. A previously established diagnosis of an active solid or hematologic malignancy.
6. A previously established diagnosis of untreated osteoporosis. For the purpose of this study, osteoporosis is defined as a dual-energy X-ray absorptiometry (DEXA) scan obtained within 2 years of screening demonstrating a hip or spine bone mineral density T score less than or equal to -2.5 in men or greater than or equal to 50 in postmenopausal women.
7. A previously established diagnosis of untreated osteopenia with a high fracture risk. For the purpose of this study, osteopenia is defined as a DEXA scan obtained within 2 years of screening demonstrating a hip or spine bone mineral density T score < -1 and > -2.5 in men or greater than or equal to 50 in postmenopausal women. For the purpose of this study, a high fracture risk is defined as a fracture risk assessment tool (FRAX) 10-year risk of major osteoporotic fracture > 20%, or a FRAX 10-year risk of hip fracture > 3%.
8. A previously established diagnosis of diabetes mellitus or a fasting blood glucose level greater than or equal to 125 mg/dL at the time of screening. For patients without a previously established diagnosis of diabetes mellitus and a fasting blood glucose level < 125 mg/dL at the time of screening, no additional screening tests (e.g., HbA1c or oral glucose tolerance test) will be performed. A history of glucocorticoid-induced hyperglycemia that is not present at the time of screening in the absence of treatment will not be considered an exclusion criterion.
9. Cancer chemotherapy within the 5 years prior to screening.
10. Surgery requiring general anesthesia in the 8 weeks prior to screening.
11. History of an infection requiring IV antibiotics in the 30 days prior to screening.
12. A positive test for HIV or hepatitis A, B, or C virus infection.
13. A positive or indeterminate test for active or latent tuberculosis (interferon gamma release assay [IGRA]) without evidence of prior treatment.
14. History of chronic or possible latent untreated parasitic, amebic, fungal, or mycobacterial infections.
15. Use of desmopressin in the 30 days prior to screening.
16. Use of one of the following cytochrome P450 isozyme (CYP) 3A4 inducers in the 30 days prior to screening: nafcillin, rifabutin, rifampin, St. John s wort, or troglitazone.
17. Use of one of the following CYP3A4 inhibitors in the 30 days prior to screening: clarithromycin, itraconazole, or ketoconazole.
18. Use of belimumab or rituximab within the past 180 days.
19. Vaccination within the past 30 days.
20. Pregnancy, current or in the 90 days prior to screening.
21. Currently breastfeeding.
22. Any electrocardiogram (ECG) abnormality that is clinically significant.
23. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Laboratory evaluations that will be used to establish eligibility are listed in sections 6 and 7, below. For exclusion criteria that involve previously established diagnoses, such as active malignancy, osteoporosis, or diabetes mellitus, any previously obtained diagnostic studies will be considered, but diagnostic testing for the sole purpose of establishing eligibility will not be performed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Franco, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Human data generated in this study will be shared for future research as follows:
  * De-identified data in an NIH-funded or approved public repository. Gene expression data will be made available through the Gene Expression Omnibus and Sequence Read Archive repositories.
  * De-identified data in public repositories.
  * Identifiable data in the Biomedical Translational Research Information System (BTRIS, automatic for activities in the CC) or the Genomic Research Integration System (GRIS).
  * De-identified or identifiable data with approved outside collaborators under appropriate agreements.
  * In publications and/or public presentations.

REFERENCES:
- [Background] Franco LM, Gadkari M, Howe KN, Sun J, Kardava L, Kumar P, Kumari S, Hu Z, Fraser IDC, Moir S, Tsang JS, Germain RN. Immune regulation by glucocorticoids can be linked to cell type-dependent transcriptional responses. J Exp Med. 2019 Feb 4;216(2):384-406. doi: 10.1084/jem.20180595. Epub 2019 Jan 23. PMID 30674564
- [Background] Cain DW, Cidlowski JA. Immune regulation by glucocorticoids. Nat Rev Immunol. 2017 Apr;17(4):233-247. doi: 10.1038/nri.2017.1. Epub 2017 Feb 13. PMID 28192415
- [Background] Stahn C, Buttgereit F. Genomic and nongenomic effects of glucocorticoids. Nat Clin Pract Rheumatol. 2008 Oct;4(10):525-33. doi: 10.1038/ncprheum0898. Epub 2008 Sep 2. PMID 18762788
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-AR-0032.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: of the 47 participants consented, six were screen failure so were not randomized to any arm in the study.
Period: Overall Study
Arm/Group | Group A: Glucocorticoids 1 mg/kg Dose | Group B: Glucocorticoids 250 mg Dose
Started | 20 | 21
Completed | 20 | 20
Not Completed | 0 | 1
Not completed — Unable to obtain specimen | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Glucocorticoids 1 mg/kg Dose | Group B: Glucocorticoids 250 mg Dose | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 11 | 13 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 6 | 10 | 16
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of SLE Patients That Were Sampled for RNA-seq Differential Expression Analysis (Biological Replicates)
Description: Number of of SLE patients that were sampled for RNA-seq differential gene expression analysis in glucocorticoid-treated immune cells. The analysis employed a cutoff value of < 5% false-discovery rate (FDR) to select the transcripts that were considered differentially expressed at each time point. The resulting gene lists were contrasted to determine which genes were uniquely differentially expressed in different cell types.
Time Frame: 2 hours and 4 hours post infusion
Population: Participants who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Glucocorticoids 1 mg/kg Dose | Group B: Glucocorticoids 250 mg Dose
Number analyzed (Participants) | 20 | 20
Participants
  2 hours post infusion | 20 | 20
  4 hours post infusion | 20 | 20

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Group A: Glucocorticoids 1 mg/kg Dose | Group B: Glucocorticoids 250 mg Dose
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 7/20 | 7/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Glucocorticoids 1 mg/kg Dose (N=20) | Group B: Glucocorticoids 250 mg Dose (N=21)
Palpitations (Cardiac disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Thirst (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 4 | 2
Tearfulness (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT04233164/Prot_SAP_000.pdf